CLINICAL TRIAL: NCT06877494
Title: Exploratory Study on the Effects of Fish Oil Supplements on Choroidal Thickness and Blood Flow Perfusion in Children and Adolescents
Brief Title: the Effects of Fish Oil Supplements on Choroidal Thickness and Blood Flow Perfusion in Children and Adolescents
Acronym: FOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YFZXYDK20240115
Record Dates: First submitted 2025-03-11; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-07

CONDITIONS: Fish Oils
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- no-treatment control group (No Intervention): No intervention measures are applied
- fish oil supplement group (Experimental): Twice a day, with one dose of DHA 300mg: EPA 60mg, for a continuous intervention of 90 days
  Interventions: Dietary Supplement: fish oil

INTERVENTIONS:
Dietary Supplement: fish oil — Twice a day, with one dose of DHA 300mg: EPA 60mg, for a continuous intervention of 90 days
  Arms: fish oil supplement group

SUMMARY:
The goal of this clinical trial is to test the effect of fish oil supplement in terms of vision in children and adolescents. The main question it aims to answer is:

the differences in changes of choroidal thickness, choroidal blood flow, axial length, and visual acuity between the intervention group and the control group Participants will take the fish oil supplement. a baseline examination will be conducted, followed by follow-up visits at 15, 30, and 90 days after the start of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 6-9 years old, gender unspecified;
2. Equivalent spherical power after unilateral cycloplegic eye ranging from 0.75D to -0.5D, with astigmatism not exceeding 1.5D;
3. Best corrected visual acuity of at least 1.0;
4. Ability to sign an informed consent form with the presence and understanding of a parent or guardian.

Exclusion Criteria:

1. Allergy or intolerance to ω-3 PUFAs or cycloplegics;
2. Strabismus, history of eye surgery (including strabismus correction surgery), other eye diseases, or systemic diseases;
3. Currently using myopia prevention measures.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2024-07-21 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Axial length | 15±2 days, 30±2 days, and 90±2 days
  the change of axial length

SECONDARY OUTCOMES:
change in equivalent spherical | 15±2 days, 30±2 days, and 90±2 days
  change in equivalent spherical in both eyes

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China